CLINICAL TRIAL: NCT00560638
Title: A Double-Masked, Randomized, Placebo-Controlled Study of Loteprednol Etabonate Ophthalmic Suspension, 0.5% for the Treatment of Dry Eye Used Either TID or QID for a 2 Week Period
Brief Title: Loteprednol Etabonate Opthalmic Suspension for the Treatment of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Tuyen Ong, MD, Bausch & Lomb Incorporated
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 439
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Loteprednol Etabonate TID (Experimental): loteprednol etabonate ophthalmic suspension, 0.5%, TID
  Interventions: Drug: loteprednol etabonate ophthalmic suspension, 0.5%
- Loteprednol Etabonate QID (Experimental): loteprednol etabonate ophthalmic suspension, 0.5%, QID
  Interventions: Drug: loteprednol etabonate ophthalmic suspension, 0.5%
- Vehicle (Placebo Comparator): vehicle of loteprednol etabonate
  Interventions: Drug: vehicle of loteprednol etabonate

INTERVENTIONS:
Drug: loteprednol etabonate ophthalmic suspension, 0.5% — TID
  Other Names: Lotemax
  Arms: Loteprednol Etabonate TID
Drug: loteprednol etabonate ophthalmic suspension, 0.5% — QID
  Other Names: Lotemax
  Arms: Loteprednol Etabonate QID
Drug: vehicle of loteprednol etabonate — TID or BID according to the randomization
  Arms: Vehicle

SUMMARY:
This was a single-center, randomized, double-masked, placebo-controlled, parallel-group, 4-visit, CAE (Controlled Adverse Environment) study lasting approximately 4 weeks. Subjects were randomized to receive loteprednol etabonate ophthalmic suspension, 0.5% or placebo (vehicle of loteprednol etabonate ophthalmic suspension, 0.5%) and instructed to dose bilaterally either TID or QID according to randomization.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age or older
* able and willing to follow instructions, including participation in study assessments and able be present for the required study visits for the duration of the study
* If female and of childbearing potential, were not pregnant, nursing, or planning a pregnancy. Women of childbearing potential were required to have a negative urine pregnancy test at the pre-screen visit and had to agree to use an acceptable method of mechanical or hormonal contraceptive for the duration of the study
* a diagnosis of dry eye
* a history of intermittent or regular artificial tear use within the past 3 months
* best corrected visual acuity (BCVA) of +0.7 or better assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in one or both eyes
* a fluorescein staining score of ≥ 1+ in at least one region in at least one eye at Visit 1 and before CAE exposure at Visits 2 and 3 OR a fluorescein staining score of ≥ 1+ in at least one region in at least one eye at Visit 1 and before CAE exposure at Visits 2 and 3 with a conjunctival redness score of ≥ 1.5+ at Visit 1 and before CAE exposure at Visits 2 and 3 in at least one eye
* Demonstrated a response when exposed to the CAE at Visits 2 and 3

Exclusion Criteria:

* clinically significant blepharitis or Meibomian Gland Dysfunction (MGD) or lid margin inflammation, particularly if systemic or topical medications were currently being used to treat any of these diagnoses
* diagnosed with an on-going ocular infection (bacterial, viral, or fungal), or active ocular inflammation (e.g. follicular conjunctivitis), or preauricular lymphadenopathy, particularly if systemic or topical medications were currently being used to treat any of these diagnoses
* Reported an ocular discomfort score of 4+ in both eyes at time 0 of CAE exposure at Visits 2 or 3
* Wore contact lenses and refused to remove them for the duration of the study
* previous laser in situ keratomileusis (LASIK) surgery
* currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs and could not discontinue these medications for the duration of the study
* presently taking any medication known to cause ocular drying that had not been a stable dose for at least 30 days
* currently taking oral antihistamines that could not be discontinued during the study
* a systemic disease, uncontrolled medical condition that in the opinion of the investigator could interfere with study measurements or subject compliance
* received another experimental drug or device within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Ocular discomfort during CAE exposure | during CAE exposure
Corneal and conjunctival staining and conjunctival redness | After CAE exposure

SECONDARY OUTCOMES:
Corneal and conjunctival staining and conjunctival redness | before CAE exposure
Blink rate, Tear film break-up time (TFBUT), and Ocular Protection Index (OPI) | before after CAE exposure
Ocular discomfort | collected in patient diaries

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Ophthalmic Research Associates, Inc.
Locations (1):
- Ophthalmic Research Associates, Andover, Massachusetts, United States